CLINICAL TRIAL: NCT05471687
Title: Evaluation of the Functional Impact of Coronary Stenoses in Diabetics by Spectral CT
Acronym: EURECAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0931
Record Dates: First submitted 2022-06-30; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Coronary Stenosis; Diabetic
Keywords: coronary stenosis; diabetics; coronary calcium score; spectral CT
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with CAC ≥ 300 three years ago (Experimental): Patients with CAC ≥ 300 three years ago with the need for repeat screening. Adult asymptomatic diabetic patients whose risk of ischemic complications is considered major in primary prevention due to a calcium score >300 AU and requiring iterative screening for IMS recommended every 3 at 5 years.
  Interventions: Device: dual-energy dual-layer spectral scanner; Drug: Stress protocol with adenosin during dual-energy dual-layer spectral scanner
- Patients with CAC between 200-299 three years ago (Experimental): Patients with CAC between 200 and 299 three years ago, with the need for a reassessment of their cardiovascular risk.
  Adult asymptomatic diabetic patients whose risk of ischemic complications is considered major in primary prevention due to a calcium score that has become pathological > 300 AU during the reassessment of their cardiovascular risk.
  Interventions: Device: dual-energy dual-layer spectral scanner; Drug: Stress protocol with adenosin during dual-energy dual-layer spectral scanner
- Patients with a recent positive scintigraphy (< three months) (Experimental): Patients with a recent positive scintigraphy (< three months) requiring coronary angiography Stable symptomatic diabetic adult patients, suspected of coronary insufficiency in whom the assessment included a positive scintigraphy with indication of coronary angiography in the perspective of revascularization.
  Interventions: Device: dual-energy dual-layer spectral scanner; Drug: Stress protocol with adenosin during dual-energy dual-layer spectral scanner

INTERVENTIONS:
Device: dual-energy dual-layer spectral scanner — Realization of dual-energy dual-layer spectral scanner with stress protocol
Drug: Stress protocol with adenosin during dual-energy dual-layer spectral scanner — Injection of intraveinous adenosin dose 0.78 mg/kg during dual-energy dual-layer spectral scanner

SUMMARY:
The optimal screening methods for coronary insufficiency, a frequent and pejorative complication in diabetics, are subject to debate, particularly in situations of silent myocardial ischemia. The contemporary strategy consists of pre-selecting asymptomatic patients at very high cardiovascular (CV) risk by performing a coronary calcium score. If this is found to be high >300 AU (Agatston units), the patient is suspected of being at high risk of silent myocardial ischemia (SMI), and the assessment is completed to exclude the presence of coronary artery disease likely to benefit from revascularization.

The complementary evaluation consists in evaluating the myocardial perfusion to judge the perfusion repercussions. The most common examination to date is myocardial scintigraphy, because stress tests are too frequently submaximal in diabetics. However, the reproducibility of scintigraphy is controversial and their sensitivity and specificity are debated in this indication.

This problem is similar in stable symptomatic coronary diabetic patients for whom an indication for functional examinations is justified.

The double-energy double-layer spectral scanner (SDEDC) could now become a relevant tool in this field, since it can combine not only anatomical data (identification of coronary stenosis) but also functional data (myocardial perfusion) during a stress protocol. thanks to the spectral images which make it possible to measure the tissue concentration of intramyocardial iodine downstream of the considered stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged man ≥50 years old or woman aged ≥55 years old, (age difference justified for established menopause which increases the CV risk and to avoid the risk of CT scan during pregnancy)
* Diabetic (type 1 or type 2 or type 3):
* Asymptomatic, falling within the scope of screening for silent myocardial ischemia and having a CAC > 300 AU or
* Symptomatic on the coronary level, within the framework of the evaluation of symptomatic coronary insufficiency with positive myocardial scintigraphy.
* Patient having agreed to participate in the study and signed a written informed consent
* Patient affiliated to a social security scheme or similar

Exclusion Criteria:

Drug intolerance (adenosine, and/or contrast product used (Iomeron))

Related to iodine injection:

* History of major immediate or delayed skin reaction + hypersensitivity to the active substance or to any of the excipients
* Renal failure with GFR < 45 ml/min -
* Known autonomic goiter with risk of thyrotoxicosis
* No suspension of the biguanide the same day of the examination (and resumed 48 hours later)

Linked to the injection of adenosine and regadenoson (Cf SPC Adenoscan combination with dipyridamole)

* 2nd or 3rd degree BAV not fitted, sinus dysfunction not fitted,
* Long QT syndrome,
* Decompensated heart failure,
* Unstable angina / Acute coronary syndrome / ATCD IDM less than a year old
* BP > 1800 mmHg < 100 mmHg
* Known stenosis of the common trunk (left),
* Tight heart valve stenosis.
* Uncorrected hypovolemia,
* Chronic obstructive pulmonary disease with clinical bronchospasm (e.g. bronchial asthma)
* Comitiality
* No suspension of dipyridamole (during the 48 hours before the examination)
* Severe hypotension
* Consumption of coffee, tobacco, tea, cola, banana, chocolate consumed before the examination (usual instructions in the event of myocardial stress protocol by adenosine agonist during the scintigraphy)
* Contraindication to adenosine: severe hypotension

Related to scanner performance

* patient unable to maintain apnea.
* Calcium score > 500 on the common trunk
* Temporary suspension of bradycardia or anti-anginal on the day of the examination (beta blocker, calcium channel blocker) not carried out.

Related to the patient's context

* Person unable to express their consent.
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Identification of tight coronary stenoses justifying coronary angiography | Measured at day 0
  An anomaly considered significant corresponds to:
  * the presence of coronary stenosis >50% with significant hypoperfusion or stenosis > 75% by spectral CT (SDEDC)
  * of a significant hypoperfusion on myocardial scintigraphy (SPECT)
  Reading Committee: Creation of a blind review committee for myocardial SPECT scans and the SDEDC spectral scanner, without knowledge of the coronary angiography data or the other perfusion examination for statistical comparison.

SECONDARY OUTCOMES:
Identification of tight coronary stenoses justifying a coronary angiography including a measurement of the Fractional Flow Reserve (FFR) | Measured at day 0
  An anomaly considered significant corresponds to:
  * the presence of coronary stenosis >50% with significant hypoperfusion or stenosis > 75% by spectral CT (SDEDC)
  * of a significant hypoperfusion on myocardial scintigraphy (SPECT)
  Reading Committee: Creation of a blind review committee for myocardial SPECT scans and the SDEDC spectral scanner, without knowledge of the coronary angiography data or the other perfusion examination for statistical comparison.
Sensitivity and specificity of the study | Measured at day 0
  Sensitivity and specificity of the study of the perfusion at rest during the SDEDC: 1 to 1 comparison of the data of the SDEC at rest (stenosis and perfusion) with the FFR; with the sensitivities and specificities of SDEDC perfusion to stress; with SPECT scintigraphy under stress.
  Reading Committee: Creation of a blind review committee for myocardial SPECT scans and the SDEDC spectral scanner, without knowledge of the coronary angiography data or the other perfusion examination for statistical comparison.
Proportion of mismatches in diabetics and their predisposing factors | Measured at day 0
  Proportion of mismatches in diabetics and their predisposing factors by identifying tissue perfusion defects (SPECT or SDEDC positive) in patients with a coronary network without angiographically tight stenosis (negative coronarography).
  Reading Committee: Creation of a blind review committee for myocardial SPECT scans and the SDEDC spectral scanner, without knowledge of the coronary angiography data or the other perfusion examination for statistical comparison.
Collection of the subjective assessment of the 2 examinations (SDEDC and myocardial scintigraphy) | Measured at day 1 and 2
  Collection of the subjective assessment of the 2 examinations (SDEDC and myocardial scintigraphy) by the patients using a satisfaction questionnaire by telephone call.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France